CLINICAL TRIAL: NCT04476368
Title: Effect of Yoga in Pregnancy on Cardiovascular and Respiratory Adaptation to Acute Psychological Challenge
Brief Title: Effect of Yoga in Pregnancy on Cardio-respiratory Adaptation to Challenge
Acronym: YOGADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, professor, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0120-575/2018/5
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Yoga; Pregnancy; Autonomic Nervous System
Keywords: yoga; pregnancy; cardiorespiratory synchronisation; hearth rate variability
MeSH Terms: interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Experimental): Participants in yoga group will be recruited during prenatal yoga classes at two locations: Maribor and Ljubljana. Women will be instructed to attend one class per week. Classes will consist of pregnancy-adapted yoga practices according to the system Yoga in Daily Life. They will be 90 min in duration and will consist of initial relaxation (10 to 15 min), followed by yoga postures (asanas) and stretching exercises (45 to 60 min), and final breathing (pranayama), concentration (dharana), and meditation (dhyana) techniques (20 to 30 min). Two certified yoga instructors will lead yoga classes. Measurements will be performed before and after yoga session.
  Interventions: Other: weekly yoga classes
- control (Active Comparator): Control group will consist of healthy pregnant women attending regular prenatal visits at the departments of perinatology of the university medical centers Maribor and Ljubljana. Only women not attending any formal prenatal exercise program will be offered entrance in the study. Measurements in this group will be performed before and after a 20-30 minute walk.
  Interventions: Other: walk

INTERVENTIONS:
Other: weekly yoga classes — Weekly 90 min pregnancy-adapted yoga classes lead by certified yoga instructors.
  Arms: yoga
Other: walk — 20-30 min easy walking
  Arms: control

SUMMARY:
Yoga has received considerable attention for its potential therapeutic benefits over the past decades and it gradually became object of scientific scrutiny. There is currently extensive literature supporting its use as a non-pharmacological tool for managing a variety of medical problems. A few studies have also explored potential beneficial effects of practising yoga during pregnancy on maternal and neonatal outcomes. An association between prenatal yoga and decreased incidence of fetal growth restriction, preterm delivery, and labor abnormalities resulting in operative delivery have been reported.

Exact mechanisms by which yoga could improve perinatal outcomes have not been elucidated yet. One of such mechanisms could be the positive effect of yoga on autonomic nervous system (ANS). Maternal cardiovascular system undergoes profound changes during pregnancy and ANS plays a central role in adaptation to pregnancy-related hemodynamic changes. Increase in peripheral vascular resistance that characterises hypertensive disorders in pregnancy with fetal growth restriction is mediated by substantial increase in sympathetic vasoconstrictor activity. Effects of yoga on ANS outside of pregnancy have already been investigated in several studies. Heart rate variability (HRV) indices, used as a one of proxy measures for ANS activity, showed significant shifts towards parasympathetic dominance following yoga sessions. Another objective means of assessing ANS activity is measurement of phase synchronisation between cardiovascular and respiratory systems following acute challenge. The higher the cardiorespiratory synchronisation after acute challenge is, the higher is the ability of ANS to flexibly adapt to challenge.

The objectives of the study are:

I. To examine whether there is a short-term shift in autonomic balance to the parasympathetic branch of the ANS and ability of the cardiovascular and respiratory respiratory systems to flexibly adapt to acute psychological challenge following sessions in pregnancy.

II. To investigate potential long- term effects of yoga practice during pregnancy on HRV and cardio-respiratory synchronisation following acute psychological challenge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women with singleton pregnancies.

Exclusion Criteria:

* Multiple pregnancies
* Cardiovascular disease (including hypertension and arrhythmias)
* Taking medications that would affect heart rate or blood pressure
* Psychiatric disorders
* Epilepsy
* Kidney disease
* Liver disease
* Known fetal anomaly
* Autoimmune disorders
* Thyroid disease
* Diabetes mellitus
* Alcohol/drug abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in cardio-respiratory phase synchronisation index | Change in cardio-respiratory phase synchronisation index from baseline (measured up to 30 minutes before yoga class/walk) to the end of exercise (measured up to 30 minutes after the end of yoga class/walk)
  Cardio-respiratory phase synchronisation index measures synchronisation between the cardiovascular and respiratory system following acute psychological challenge. It's value is between 0 (no synchronisation) and 1 (complete synchronisation). The higher the value, the higher the ability of cardiovascular and respiratory systems to flexibly adapt to challenge (standardised memory task).
Change in LF/HF HRV ratio. | Change in LF/HF HRV ratio from baseline (measured up to 30 minutes before yoga class/walk) to the end of exercise (measured up to 30 minutes after the end of yoga class/walk).
  For frequency related HRV indices, we will run an autoregressive spectral analysis using Burg's algorithm (model order 24) after resampling and removing the trend of 2nd order. Low frequency (LF) will be defined as 0.04 - 0.15 Hz, high frequency (HF) will be defined as 0.15 - 0.40 Hz. The higher the LF/HF HRV ratio, the lower the parasympathetic tone.
BRS | Change in BRS from baseline (measured up to 30 minutes before yoga class/walk) to the end of exercise (measured up to 30 minutes after the end of yoga class/walk).
  The sequence technique will be used for the assessment of baroreceptor sensitivity (BRS). This technique is based on identifying consecutive cardiac beats in which an increase in systolic blood pressure is accompanied by an increase in heart rate, or in which a decrease in systolic blood pressure is accompanied by a decrease in heart rate. The regression line between the systolic blood pressure and heart rate produces an estimate of BRS. The higher the BRS, the higher the parasympathetic tone.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - UMC Ljubljana, Ljubljana
  - UMC Maribor, Maribor

IPD SHARING:
Plan to Share IPD: Yes